CLINICAL TRIAL: NCT05636137
Title: Analysis of Internet Addiction, Musculoskeletal Pain and Body Awareness in High School Students
Status: Enrolling by invitation | Type: Observational
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Burcu Camcıoğlu Yılmaz, PT, PhD, Muğla Sıtkı Koçman University
Other Study IDs: MEB1
Record Dates: First submitted 2022-11-23; First posted 2022-12-05 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-05

CONDITIONS: Healthy
Keywords: Internet Addiction; Musculoskeletal Pain; Body Awareness; High School; Students
MeSH Terms: conditions — Internet Addiction Disorder; Musculoskeletal Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- High School Students: The sample of the study consists of high school students who do not have mental disabilities that will prevent them from understanding and answering the questions, aged 15-18 and volunteer to participate in the study, have internet at home and have an individual device that provides internet access.
  Interventions: Other: Survey application

INTERVENTIONS:
Other: Survey application — Researchers will go to the designated high schools and meet face-to-face with the responsible/guidance teachers at the school. The research will be explained to the students by going to the classrooms with the teachers, and they will be asked to fill in the consent forms of the parents and themselves. Students will be given 5 days to explain the work to their families and bring their signed consent forms. Students who bring consent forms, meet the criteria for participation in the study, and volunteer will be included in the study. Evaluation forms and questionnaires will be explained to the students included in the study by a designated researcher and they will be asked to fill them in under the supervision of the researcher. The completed evaluation form and questionnaires will be collected by a researcher in a sealed envelope.

SUMMARY:
The study will investigate internet addiction, musculoskeletal pain and body awareness in high school students.

DETAILED DESCRIPTION:
Internet addiction is generally defined as not being able to prevent excessive use of the internet, the time spent on other occupations is not as valuable as the internet, excessive irritability and aggressive behavior when deprived.This situation brings with it musculoskeletal pain. Pain in the musculoskeletal system can cause a decrease in body awareness.Long periods of time spent in front of the computer, the use of non-ergonomic tables and chairs affect body awareness by causing deterioration of posture. There are several studies in literature investigating internet addiction and pain, however internet addiction, body awareness and musculoskeletal system problems of high school students have not been investigated yet. In present study, internet addiction, body awareness and musculoskeletal problems will be investigated in high school students.

ELIGIBILITY:
Inclusion Criteria:

* Not having a mental disability that will prevent them from understanding and answering the questions
* 15-18 years old
* Having internet at home
* Volunteering to participate in the study
* Having an individual device that provides internet access

Exclusion Criteria:

* No family approval
* Having an orthopedic, musculoskeletal or neurological disease that will affect body awareness and musculoskeletal system.

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Students will be included from high schools in Muğla that do not provide technical and vocational education. 213 students who met the criteria for participation in the study and volunteered will be included in the study. Students will be between the ages of 15-18.
Sampling Method: Non-Probability Sample
Enrollment: 213 (Estimated)
Dates: Start 2025-07-24 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Internet Addiction Scale | 5-10 minutes
  This questionnaire consists of 20 statements. After reading each statement carefully, based upon the 5-point Likert scale. Total scores that range from 0 to 30 points are considered to reflect a normal level of Internet usage; scores of 31 to 49 indicate the presence of a mild level of Internet addiction; 50 to 79 reflect the presence of a moderate level; and scores of 80 to 100 indicate a severe dependence upon the Internet
Body Awareness Questionarre | 5-10 minutes
  It is a scale that questions the level of physiological, psychological, emotional and social awareness of the individual, the differences between sleep disorder, being sick and not being sick, bodily and mental reactions in specific situations related to body awareness, and the level of estimation.
Cornell Musculoskeletal Discomfort Questionnaires | 5-10 minutes
  The frequency and severity of the discomfort they have experienced are presented to the participants as options, and they are expected to answer the option appropriate for their situation according to the last week.

CONTACTS AND LOCATIONS:
Overall Officials: Burcu Camcıoğlu Yılmaz, PT,PhD, Study Director — Muğla Sıtkı Koçman University; Merve Gürkan, MSc.Student, Principal Investigator — Muğla Sıtkı Koçman University
Locations (1):
- Mugla Sitki Kocman University Faculty of Health Sciences, Muğla, Menteşe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sinkkonen HM, Puhakka H, Merilainen M. Internet use and addiction among Finnish adolescents (15-19 years). J Adolesc. 2014 Feb;37(2):123-31. doi: 10.1016/j.adolescence.2013.11.008. Epub 2013 Dec 10. PMID 24439618
- [Background] Sung J, Lee J, Noh HM, Park YS, Ahn EJ. Associations between the Risk of Internet Addiction and Problem Behaviors among Korean Adolescents. Korean J Fam Med. 2013 Mar;34(2):115-22. doi: 10.4082/kjfm.2013.34.2.115. Epub 2013 Mar 20. PMID 23560210
- [Background] Kim Y, Park JY, Kim SB, Jung IK, Lim YS, Kim JH. The effects of Internet addiction on the lifestyle and dietary behavior of Korean adolescents. Nutr Res Pract. 2010 Feb;4(1):51-7. doi: 10.4162/nrp.2010.4.1.51. Epub 2010 Feb 24. PMID 20198209
- [Background] Cao H, Sun Y, Wan Y, Hao J, Tao F. Problematic Internet use in Chinese adolescents and its relation to psychosomatic symptoms and life satisfaction. BMC Public Health. 2011 Oct 14;11:802. doi: 10.1186/1471-2458-11-802. PMID 21995654
- [Background] Harman JP, Hansen CE, Cochran ME, Lindsey CR. Liar, liar: internet faking but not frequency of use affects social skills, self-esteem, social anxiety, and aggression. Cyberpsychol Behav. 2005 Feb;8(1):1-6. doi: 10.1089/cpb.2005.8.1. PMID 15738687
- [Background] Paananen MV, Auvinen JP, Taimela SP, Tammelin TH, Kantomaa MT, Ebeling HE, Taanila AM, Zitting PJ, Karppinen JI. Psychosocial, mechanical, and metabolic factors in adolescents' musculoskeletal pain in multiple locations: a cross-sectional study. Eur J Pain. 2010 Apr;14(4):395-401. doi: 10.1016/j.ejpain.2009.06.003. Epub 2009 Jul 28. PMID 19640750
- [Background] Mehling WE, Gopisetty V, Daubenmier J, Price CJ, Hecht FM, Stewart A. Body awareness: construct and self-report measures. PLoS One. 2009;4(5):e5614. doi: 10.1371/journal.pone.0005614. Epub 2009 May 19. PMID 19440300
- [Background] Baas LS, Beery TA, Allen G, Wizer M, Wagoner LE. An exploratory study of body awareness in persons with heart failure treated medically or with transplantation. J Cardiovasc Nurs. 2004 Jan-Feb;19(1):32-40. doi: 10.1097/00005082-200401000-00007. PMID 14994780
- [Background] Barron CR, Foxall MJ, Houfek JF. Coping style and women's participation in breast and gynecological screening. Health Care Women Int. 2005 Mar;26(3):247-61. doi: 10.1080/07399330590917807. PMID 15804696
- [Background] Bekker MH, Croon MA, van Balkom EG, Vermee JB. Predicting individual differences in autonomy-connectedness: the role of body awareness, alexithymia, and assertiveness. J Clin Psychol. 2008 Jun;64(6):747-65. doi: 10.1002/jclp.20486. PMID 18425792
- [Background] Boyle CA, Sayers SP, Jensen BE, Headley SA, Manos TM. The effects of yoga training and a single bout of yoga on delayed onset muscle soreness in the lower extremity. J Strength Cond Res. 2004 Nov;18(4):723-9. doi: 10.1519/14723.1. PMID 15574074
- [Background] Erdinc O, Hot K, Ozkaya M. Turkish version of the Cornell Musculoskeletal Discomfort Questionnaire: cross-cultural adaptation and validation. Work. 2011;39(3):251-60. doi: 10.3233/WOR-2011-1173. PMID 21709361
- See also: Internet Addiction and Its Treatment — http://dergipark.org.tr/tr/pub/pgy/issue/11166/133473
- See also: Household Information Technologies (IT) Usage Survey — http://data.tuik.gov.tr/Bulten/Index?p=Hanehalki-Bilisim-Teknolojileri-(BT)-Kullanim-Arastirmasi-2022-45587
- See also: A RESEARCH ON THE USE OF SOCIAL NETWORKS OF UNIVERSITY STUDENTS — http://dergipark.org.tr/tr/pub/usakjhs/issue/13534/163818
- See also: Examining the Relationship Between Cyberbullying and Problematic Internet Use and Risky Internet Behavior — http://dergipark.org.tr/tr/pub/tebd/issue/32959/328896
- See also: Effects of internet use and internet addiction in line with media addiction theory — http://search.trdizin.gov.tr/yayin/detay/96714/
- See also: Internet Addiction: A Current Review — http://dergipark.org.tr/tr/download/article-file/222170
- See also: THE EFFECT OF SCREEN BASED ACTIVITIES ON HAMSTRING MUSCLE LENGTH, REACTION TİME AND BODY MASS INDEX IN ADOLESANS — http://dergipark.org.tr/tr/download/article-file/53593
- See also: The Effect of Technology Addiction on Posture and Body Awareness in School Age Children — http://dergipark.org.tr/tr/download/article-file/791897
- See also: Üniversite Öğrencilerinin Kas İskelet Sistemi Rahatsızlıkları ile Fiziksel Aktivite Düzeyi ve İnternet Bağımlılığı Arasındaki İlişkinin İncelenmesi — http://dergipark.org.tr/tr/download/article-file/1979865
- See also: Internet addiction and sleep disturbance symptoms among Turkish high school students — https://link.springer.com/article/10.1111/sbr.12022
- See also: The Study Of Validity And Reliability Of The Social Media Addiction Scale Short Form For Adolescents — http://dergipark.org.tr/tr/download/article-file/320071
- See also: TURKISH VERSION OF BODY AWARENESS QUESTIONARRE: VALIDITY AND RELIABILITY STUDY — http://acikbilim.yok.gov.tr/handle/20.500.12812/222691
- See also: Inner body and outward appearance- the relationship between orientation toward outward appearance, body awareness and symptom perception — http://research.tilburguniversity.edu/en/publications/inner-body-and-outward-appearance-the-relationship-between-orient